CLINICAL TRIAL: NCT06830278
Title: The Efficacy of a New Sexual Violence Primary Prevention Program for Adolescents: A Cluster Randomized Trial of the Stand Up Now Against Sexual Violence (SUN) Program
Brief Title: The Efficacy of the SUN Program in Adolescents
Acronym: SUN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: University of Coimbra (Other); Aveiro University (Other); Faculty of Medicine of the University of Porto (Unknown); Foundation for Science and Technology, Portugal (Other); Center for Psychology at the University of Porto, Portugal (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SUN-2024-EC
Record Dates: First submitted 2024-12-23; First posted 2025-02-17 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Sexual Violence
Keywords: Adolescents; Bystanders; Prevention; Psychoeducation; Sexual Violence; School settings; Skills training

STUDY DESIGN:
Intervention Model Description: Participants in the control groups take part in the scheduled in-person school activities, as usual. Participants in the intervention group take part in the in-person sessions of the SUN Program. This is a parallel design, so participants are part of the same group for the duration of the entire study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The students in the control cluster continue scheduled school activities as usual.
- Experimental group (Experimental): Participants in the intervention cluster take part in the SUN Program.
  Interventions: Behavioral: The SUN Program

INTERVENTIONS:
Behavioral: The SUN Program — The SUN Program is a manualized bystander program for high-school adolescents. The program includes ten 50-to-60 minute weekly sessions. The central contents of the program include sexual and reproductive rights, sexual violence throughout the lifespan in different contexts, bystander attitudes and behaviors, and empathy. Every session includes psychoeducation components as well as skills-training moments. The sessions must be delivered by two psychologists with supervision.
  Session contents are divided as following:
  Session 1: Introduction to sexual violence and sexual rights; Session 2: Sexual violence: behaviors and contexts, Session 3: Sexual consent; Session 4: Sexual violence myths; Session 5: Sexual violence in intimate relationships; Session 6: The role of the bystanders; Session 7: The bystander effect; Session 8: Bystander intervention; Session 9: Empathy; Session 10: Summary
  Arms: Experimental group

SUMMARY:
This research project will develop, deliver, and evaluate a new school-based sexual violence prevention program for high-school adolescents. The SUN program (Stand Up Now against sexual violence) aims to prevent the occurrence of sexual violence among adolescents. The program approaches sexual violence as a complex phenomenon which occurs in many contexts throughout life. This program approaches specific concepts associated with sexual violence, such as sexual consent, while acknowledging the association between this form of violence and other violent phenomena. The program uses a bystander approach to support adolescents in the development of bystander attitudes and behaviors, which can be used in situations where the risk of sexual violence may be present. These may include behaviors such as confronting someone who is trying to take advantage of another person or reporting someone who committed sexual violence. The program aims to reduce myths associated with sexual violence, to increase empathy in this context and to improve bystander skills. Program sessions will combine group discussions with skills-building exercises.

This study will apply the SUN program in school settings and compare the adolescents who will take part in the program with adolescents who will not. The study will evaluate changes in sexual violence myths, sexism, empathy, and bystander attitudes and behaviors. The authors hypothesize that by decreasing myths associated with sexual violence and sexism, and by increasing empathy in this context, the program will be able to increase the adolescents' capacity to intervene in real-world situations to prevent sexual violence (i.e., bystander attitudes and behaviors). Additionally, the programs' acceptability will be assessed through focus groups conducted with students. It is expected that this project will improve scientific knowledge regarding sexual violence prevention.

DETAILED DESCRIPTION:
Study Design, Aims and Hypotheses:

The main goal of the present project is to develop, deliver, and assess the efficacy of a new bystander primary prevention program for SV targeting high school adolescents in Portugal (the SUN Program: Stand Up Now against sexual violence).

This mixed-method study will involve a pragmatic parallel-arm cluster randomized controlled trial. The CRT will be conducted according to the following goals: 1) to assess the program's efficacy, by evaluating its ability to significantly increase bystander attitudes and behaviors, as well empathy; and to reduce SV myths and sexism; 2) to examine the extent to which any changes are maintained three, six and nine months after the program's completion (follow-up); 3) to assess mechanisms of change (i.e., to test whether the reduction of SV myths and sexism and the increase in empathy predicts increases in bystander attitudes and behaviors); 4) to investigate whether age, gender, sexual orientation and personal history of victimization influence the participants' responsivity to the program; 5) to assess the program's acceptability by conducting focus groups with adolescent participants.

Study hypothesis were designed in accordance with the research goals: Hypothesis (1) Participants in the experimental group (i.e., taking part in the SUN Program) will show significant increases over time in bystander attitudes, bystander behaviors and empathy, and decreases over time in SV myths and sexism when compared with participants in the control group; Hypothesis (2) The reductions of SV myths and sexism and the increases in empathy will predict increases in bystander attitudes and behaviors in adolescents from the experimental group; Hypothesis (3) Age, gender, sexual orientation and personal history of victimization will influence participants' responsivity to the SUN program (i.e., younger participants, participants identifying with a gender or sexual minority group, and participants with a history of previous victimization will show greater responsivity to the SUN program); This research project will be conducted according to the Consort 2010 statement: extension to cluster randomized trials and to the Standards of Evidence for Efficacy, Effectiveness, and Scale-up Research in Prevention Science.

Setting and Proposed Sample:

The sample will include adolescents from high schools in the North and Centre of Portugal, enrolled in 10th and 11th grades. A sample of adolescents was selected considering the epidemiological data showing high prevalence rates of SV in this population; the differences in sexual victimization and perpetration patterns and consequences in adolescence in comparison to childhood or adulthood; and in the fact that victimization and perpetration trajectories in adolescence may act as predictors of violence in adulthood . Additionally, authors agree that early intervention during adolescence is crucial and recent evidence suggests greater efficacy of prevention programs for older adolescents, although further research is needed to clarify the ideal timing of intervention during adolescence. Grades 10 and 11 were selected to improve adherence to follow-up evaluations (i.e., to reduce to likelihood of dropout, as high school finishes in 12th grade in Portugal and contact with students via schools after that would not be feasible). Public, vocational and private schools were contacted to ensure diversity in study settings.

A priori sample size estimation accounted for the cluster randomized trial (CRT) design, in which classes are the unit of randomization. The trial includes two parallel arms (intervention vs. control) and five assessment points (baseline, post-test, 3-, 6-, and 9-month follow-ups).

Sample Size Estimation The base sample size was calculated in G*Power 3.1 for a two-tailed t-test comparing two independent means, with α = .05, power = .80, and a standardized effect size of d = 0.30, consistent with previous school-based bystander and prevention programs. This analysis indicated that 352 participants (176 per group) are required under individual randomization.

Because randomization occurs at the class level, the sample was inflated using the design effect (DE) formula.

Assuming an average class size of m = 15 students and an intraclass correlation coefficient (ICC) = 0.03, typical for psychosocial outcomes in educational settings, the design effect equals 1.42. Adjusting for clustering increases the total required sample to approximately 500 students (≈ 250 per arm), corresponding to 34 classes (17 per arm).

To accommodate 20% expected attrition over the 9-month follow-up, the final recruitment target is approximately 600 students (≈ 40 classes, 20 per arm). This sample size provides a minimum of 80% power to detect small-to-moderate effects and is sufficient for planned moderation and mediation analyses. If cluster sizes vary substantially, the design effect will be corrected using the coefficient of variation (CV) of class size.

For the mechanism-of-change analyses, an a priori RMSEA-based power analysis (power4SEM; Wolf et al., 2013) indicated that N ≈ 550 achieves 80% power for detecting model fit differences (testing RMSEA₀ = .05 vs. RMSEA₁ = .08, α = .05). The planned CRT sample (≈ 600 participants) therefore ensures sufficient power for longitudinal structural equation modeling (SEM).

Recruitment:

The recruitment process started with a series of email and phone contacts targeting schools in the North and Center of Portugal. Schools were invited to online or in-person meetings to present the SUN Program and the research project. Response rates were recorded, as well as any stated reasons for non-participation. These meetings allowed the detailed explanation of the program sessions, the consent and assent procedures, the randomization process, and all assessments. Schools were asked to discuss their interest in participating in the project, as well as their respective feasibility conditions (e.g., number of classes available, number of students per class, gender distribution of each class, school schedules). After meeting with the interested schools, researchers evaluated interest and feasibility conditions and selected a pool of schools for inclusion in the study. After the selection of four schools, the representative from each school indicated the classes selected (based on feasibility conditions). Then, presentation sessions were conducted for students in the recruited classes and their teachers, during school hours. The aim of these sessions was to share with students and teachers the information previously communicated in the school meetings (e.g., assessments and consent/assent procedures). At the end of the presentation sessions, participants younger than 18 years were given an assent form for themselves and a consent form for one of their caregivers. Participants older than 18 years were given a consent form for themselves. These ethical procedures are in line with the schools' legal regulations. Any doubts regarding these forms were clarified in person and email contacts were provided. Only about a week after the presentation sessions did researchers collect the signed consent/assent forms, to ensure participants had enough time to make an informed decision. Recruitment was concluded once participants hand in their consent and assent forms. Participants were informed that they would later be invited for participation in focus groups. Specific assent forms were signed by students who participated in the focus groups.

Randomization:

Clusters were randomly assigned to either the SUN Program condition or the control condition in a 1:1 ratio. Randomization was conducted after the baseline assessment using a randomization software (https://www.randomizer.org/). Considering the nature of this research project (i.e., a pragmatic trial), the research team, school staff and participants were not blinded to intervention conditions.

Dropout and Retention:

This research project was designed considering particular concerns regarding the minimization of the risk of bias. To avoid non-response, school staff were asked to support the research team in the monitoring of students who respond at each assessment period and to follow-up those with missing surveys. To avoid dropouts, sessions took place during school hours, normally in the middle of the school day, without colliding with other relevant school events. Participation did not involve any financial costs or travelling. Caregivers and school staff have been involved in the dissemination of the program, to increase the community's commitment with this project.

Moreover, facilitators use a trauma-informed approach to reduce any potential negative impact of the program's discussions. As such, they are available to support participants, as well as caregivers and staff both in person and online. An email account, an anonymous online form and an Instagram profile are available in case participants want to contact facilitators or researchers outside the sessions. Thus, several procedures are in place to ensure that dropouts are minimal.

Quality Assurance:

During the implementation of this research project there will be a continuous quality assurance effort, namely focused on data monitoring. Considering the sensitivity of the contents of the SUN Program and the survey questions, data safety and monitoring measures were applied. Survey materials were revised in depth before the start of the study to ensure that all ethical requirements are fulfilled. All assessment procedures were conducted by trained psychologists and researchers with victim and offender support training. Signed consent and assent forms were stored in a secure file drawer inside a locked office, separate from paper surveys. Participant names (collected to confirm the presence in the assessment sessions) were kept in password protected files accessible only to the research team. The research team did not have participants' contact details. Any communication with the participants was ensured by the school staff, to ensure participants' privacy. Only in exceptional circumstances will participants' or research staff's contact details be shared (e.g., in a disclosure situation).

Study procedures were continuously supervised, namely concerning confidentiality, privacy, and secure maintenance of data. This supervision also included availability to support research and school staff, as well as caregivers, in case of disclosures or any need of support during the application of the research project. Finally, any incidents concerning data safety, confidentiality or participant safety will be discussed, reviewed and reported.

Ethical Standards:

This project follows the ethical standards of the Declaration of Helsinki, the Ethical Principles of Psychologists and Code of Conduct of the American Psychological Association, the Code of Ethics of the Order of Portuguese Psychologists and ethical guidelines from the Sexual Violence Research Initiative and from the World Health Organization.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents
* Enrolled in high schools in grades 10th and 11th
* Enrolled in schools of the North or Center of Portugal
* Fluent in Portuguese (spoken and written)

Exclusion Criteria:

* Presence of a serious developmental disorder, physical or mental health issue that interferes with the participation in the sessions, as reported by the caregivers or by the school staff

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Bystander attitudes | All primary outcome measures will be assessed at baseline (1 week before the first session of the SUN), post-test (1 week after the last session of the SUN), and three, six and nine months after pos-test (follow-up assessments).
  Bystander attitudes - Bystander Attitude Scale-Revised (BAS-R)
  The Bystander Attitude Scale-Revised (modified version) is a self-report survey that measures bystander attitudes using 19 items (McMahon et al., 2014). This study uses a recent adaptation of this scale into Portuguese for adolescents, using only 13 items (in preparation for publication). The scale uses several items that capture a diverse range of bystander behaviors in terms of low and high risk of violence, timing of the intervention and proactive or reactive behaviors. An item example would be: "Report a friend to the police if I heard rumors that they had forced someone to have sex". In this survey, participants are asked to rate how acceptable a behavior is for them (i.e., whether they are favorable to that behavior) on a Likert scale from 1 (not acceptable) to 5 (extremely acceptable) (McMahon et al., 2014).
Bystander behaviours - Bystander Behavior Scale-Revised (BBS-R) | All primary outcome measures will be assessed at baseline (1 week before the first session of the SUN), post-test (1 week after the last session of the SUN), and three, six and nine months after pos-test (follow-up assessments).
  The Bystander Behavior Scale-Revised (modified version) is a self-report survey similar to the BAS-R but which measures bystander behavior. Items are the same but participants are asked to report whether they have had those behaviors in the previous year (scale: "Yes", "No", "I wasn't in that situation") (McMahon et al., 2014).

SECONDARY OUTCOMES:
Empathy | All secondary outcome measures will be assessed at baseline (1 week before the first session of the SUN), post-test (1 week after the last session of the SUN), and three, six and nine months after pos-test (follow-up assessments).
  The Basic Empathy Scale-Adolescents (BES-A) is a self-report questionnaire for adolescents that evaluates empathy in its affective and cognitive dimensions (Anastácio et al., 2016; Jolliffe & Farrington, 2006). This study uses the short version adapted to the Portuguese context, which includes seven items: four for the cognitive empathy subscale and three for the affective empathy subscale (Pechorro et al., 2018). Item examples include "After I talk to a friend who is sad, I generally become sad too" (affective empathy subscale) and ''When people are feeling down, I generally can understand how they are feeling'' (cognitive empathy subscale). Answers are given according to a five-point scale, ranging from 1 = strongly disagree and 5 = strongly agree.
Sexual violence myths | All secondary outcome measures will be assessed at baseline (1 week before the first session of the SUN), post-test (1 week after the last session of the SUN), and three, six and nine months after pos-test (follow-up assessments).
  The Attitudes Toward Dating Violence Scale - Portuguese adaptation (EAVN) is a self-report questionnaire for adolescents (Price et al., 1999; Saavedra, 2010). This study uses the Sexual Violence perpetrated by Men subscale (12 items) and the Sexual Violence perpetrated by Women subscale (12 items) (Saavedra, 2010). The item "When boys are very sexually aroused, they cannot avoid having sex" is an example from the Sexual Violence perpetrated by Men subscale. The item "There is nothing wrong with a girl forcing her boyfriend to kiss her" is an example from the Sexual Violence perpetrated by Women subscale. Answers are given according to a five-point Likert scale, ranging from 1 = strongly disagree and 5 = strongly agree.
Sexism | All secondary outcome measures will be assessed at baseline (1 week before the first session of the SUN), post-test (1 week after the last session of the SUN), and three, six and nine months after pos-test (follow-up assessments).
  The Scale for Detection of Sexism in Adolescents - Escala de Detección de Sexismo en Adolescentes (DSA) is a self-report questionnaire including 26 items aimed at detecting sexism in adolescents (Fernandes, 2020; Recio, 2007). The scale includes two subscales: ten items measure benevolent sexism and 16 items measure hostile sexism (Recio et al., 2007). The item "Women are, naturally, more patient and tolerant than men." provides an example of the benevolent sexism scale". Item 2 provides an example of the hostile sexism scale: "The most adequate place for a woman is at home with her family". Answers are given according to a six-point scale, ranging from 1 = strongly disagree and 6 = strongly agree.
Social Desirability | All secondary outcome measures will be assessed at baseline (1 week before the first session of the SUN), post-test (1 week after the last session of the SUN), and three, six and nine months after pos-t (follow-up assessments).
  The Social Desirability Scale - Escala de Desejabilidade Social (EDS-20) is a self-report questionnaire developed to assess social desirability in diverse samples, including adolescents (Almiro et al., 2017). Items are answered on a dichotomous scale of "Yes" or "No". An item example would be "Have you ever taken advantage of someone?". This scale will be integrated as a covariate.

CONTACTS AND LOCATIONS:
Overall Officials: Joana Carvalho, PhD, Study Director — William James Center for Research, Department of Education and Psychology, University of Aveiro; Eunice Carmo, MSc, Principal Investigator — Center for Psychology at University of Porto
Locations (1):
- Four different schools in Porto and Aveiro districts, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torazzi E, Merelli V, Barbara G, Kustermann A, Marasciuolo L, Collini F, Cattaneo C. Similarity and Differences in Sexual Violence Against Adolescents and Adult Women: The Need to Focus on Adolescent Victims. J Pediatr Adolesc Gynecol. 2021 Jun;34(3):302-310. doi: 10.1016/j.jpag.2020.11.018. Epub 2020 Nov 28. PMID 33259887
- [Background] Piolanti A, Jouriles EN, Foran HM. Assessment of Psychosocial Programs to Prevent Sexual Violence During Adolescence: A Systematic Review and Meta-analysis. JAMA Netw Open. 2022 Nov 1;5(11):e2240895. doi: 10.1001/jamanetworkopen.2022.40895. PMID 36346627
- [Background] Panisch LS, Faulkner M, Fernandez SB, Fava NM. Exploring How Trauma Is Addressed in Sexual Education Interventions for Youth: A Scoping Review. Health Educ Behav. 2020 Dec;47(6):880-893. doi: 10.1177/1090198120954398. Epub 2020 Sep 8. PMID 32900237
- [Background] McMahon S, Allen CT, Postmus JL, McMahon SM, Peterson NA, Lowe Hoffman M. Measuring bystander attitudes and behavior to prevent sexual violence. J Am Coll Health. 2014;62(1):58-66. doi: 10.1080/07448481.2013.849258. PMID 24313697
- [Background] Gottfredson DC, Cook TD, Gardner FE, Gorman-Smith D, Howe GW, Sandler IN, Zafft KM. Standards of Evidence for Efficacy, Effectiveness, and Scale-up Research in Prevention Science: Next Generation. Prev Sci. 2015 Oct;16(7):893-926. doi: 10.1007/s11121-015-0555-x. PMID 25846268
- [Background] Carmo E, Brazao N, Carvalho J. The Primary Prevention of Sexual Violence Against Adolescents in School and Community Settings: A Scoping Review. J Sex Res. 2025 May;62(4):656-672. doi: 10.1080/00224499.2024.2367562. Epub 2024 Jun 28. PMID 38940424
- [Background] Campbell MK, Piaggio G, Elbourne DR, Altman DG; CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012 Sep 4;345:e5661. doi: 10.1136/bmj.e5661. No abstract available. PMID 22951546
- [Background] Barbara G, Albertini V, Tagi VM, Maggioni L, Gorio MC, Cattaneo C, Parazzini F, Ricci E, Buggio L, Kustermann A. Characteristics of Sexual Violence Against Adolescent Girls: A 10 Years' Retrospective Study of 731 Sexually Abused Adolescents. Int J Womens Health. 2022 Mar 3;14:311-321. doi: 10.2147/IJWH.S343935. eCollection 2022. PMID 35273451